CLINICAL TRIAL: NCT02632487
Title: Wearable Technology to Reduce Sedentary Behavior and CVD Risk in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB201501139
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Active Comparator): This group will receive 8 weeks of center-based exercise followed by recommendations to remain physically active.
  Interventions: Behavioral: Exercise
- Exercise + Non-Exercise Physical Activity (NEPA) (Experimental): This group will receive 8 weeks of center-based exercise combined with behavioral counseling and a technology intervention designed to increase daily Exercise + Non-Exercise Physical Activity (NEPA).
  Interventions: Behavioral: Exercise; Behavioral: Non-Exercise Physical Activity (NEPA)

INTERVENTIONS:
Behavioral: Exercise — Center-based walking + balance, stretching, and light resistance
Behavioral: Non-Exercise Physical Activity (NEPA) — Behavioral counseling paired with technology intervention to monitor physical activity
  Arms: Exercise + Non-Exercise Physical Activity (NEPA)

SUMMARY:
This study will evaluate the feasibility and efficacy of combining a traditional, structured exercise intervention with an innovative intervention designed to decrease sedentary behavior and increase non-exercise physical activity (NEPA).

DETAILED DESCRIPTION:
A recruitment of 40 sedentary men and women ≥ 60 years of age with elevated cardiovascular risk and follow them for 20 weeks. Participants will be randomly assigned (n = 20/group) to 1) an 8-week, twice-weekly, multi-modal, center-based exercise intervention (EX) followed by 12 additional weeks of follow-up assessment, or 2) the same intervention with participants also asked to wear a validated lightweight activity tracker on their hip during waking hours and instructed on how to reduce sedentary behavior increase NEPA within their daily routines (EX + NEPA). Evaluations will be done to 1) the extent to which EX + NEPA modifies sedentary behavior, 2) the impact of the interventions on cardiovascular risk factors, including blood pressure, exercise capacity, waist circumference, and circulating biomarkers, and 3) develop and optimize study procedures to guide the future trial.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary lifestyle, defined as <150 min/wk of moderate physical activity by CHAMPS questionnaire
* Moderate to high-risk of CHD events according to ATP-III risk classification algorithm
* Willingness to be randomized to either intervention group
* Willingness to participate in all study procedures

Exclusion Criteria:

* Failure to provide informed consent;
* Regular participation in an exercise training program within the last 3 months
* Absolute contraindication(s) to exercise training (American College of Sports Medicine guidelines)
* Office SBP > 180 mm Hg or DBP > 110 mm Hg
* Severe cardiac disease, i.e. NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina;
* Myocardial infarction or stroke within past year
* Significant cognitive impairment, i.e. known dementia or a Mini-Mental State Examination score < 24
* Progressive, degenerative neurologic disease, e.g., Parkinson's Disease, multiple sclerosis, ALS;
* Severe rheumatologic/orthopedic disease, e.g., awaiting joint replacement, active inflammatory disease
* Severe pulmonary disease, requiring either steroid pills or injections or the use of supplemental oxygen;
* Hip fracture, hip or knee replacement, or spinal surgery within past 4 months;
* Other significant co-morbid conditions that would impair ability to participate in the intervention
* Simultaneous participation in another intervention trial

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Blood pressure between the groups | 20 weeks

SECONDARY OUTCOMES:
Exercise capacity between the groups | 20 weeks
  distance on 6-minute walk test
Waist circumference between the groups | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Anton, Principal Investigator — Univesity of Florida
Locations (1):
- UF Clinical Translational Research Building, Gainesville, Florida, United States